CLINICAL TRIAL: NCT05084040
Title: Non-inferiority of Clinical Trials in Comparison With the Length of Totally Implemented Porth-a-Cath Maintenance From 60 Versus 90 Days
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2663-19
Record Dates: First submitted 2021-08-13; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Catheter Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (No Intervention): Porth-a-Cath maintenance with 60-day interval
- B (Experimental): Porth-a-Cath maintenance with 90-day interval
  Interventions: Other: 90 days interval between catheter maintenance

INTERVENTIONS:
Other: 90 days interval between catheter maintenance — Length of time between catheter maintenances extended from 60 days to 90 days
  Arms: B

SUMMARY:
Abstract: Antineoplastic therapy (AT) is one of the most used treatment modalities to fight cancer, either curatively or palliatively. There are several possible routes of administration, but the intravenous is the most used for its safe absorption and maintenance of the drug's serum level (1). Among the central catheters used in oncology, the long-term Totally Implantable (CTI) catheter is one of the most well accepted by patients and healthcare professionals. Being used in the administration of fluids, medication, parenteral nutrition or to obtain blood. Maintaining the CTI is essential to maintain its permeability, and thus, its proper functioning (2-4). The COVID-19 pandemic requires several readjustments from health institutions to ensure healthy environments for patients and less exposure to the hospital environment, one of the measures to focus on increasing the maintenance time of the ICU from 30 to 60 days. Objective: To verify the safety of increasing the maintenance interval of the Port-a-Cath catheter from 30 to 60 days through the rate of infection, obstruction, dysfunction in the infusion of solutions and blood reflux at the end of a year of follow-up. Method: This is an observational study, a single research arm, with a scheduled duration from January 2021 to August 2022 at the chemotherapy clinics of the A.C.Camargo Cancer Center. Expected results: This investigation is expected to demonstrate that maintenance with saline every 60 days does not increase obstruction or infection in patients who are in clinical follow-up compared to maintenance for 30 days.

DETAILED DESCRIPTION:
1.Patients and methods

1.1. Study design

Recruitment will take place during three months in the chemotherapy ambulatory at A.C. Camargo Cancer Center. Patients will be invited to participate in this study once they undergo maintenance of the fully implanted catheter (FIC), according to institutional routine. If the invited patient meets the inclusion and exclusion criteria defined in this study, he will respond to the financial assessment (Appendix 1). In the next step, he will be instructed to wait for the researcher to contact him to inform the next day of catheter maintenance.

After the clinical findings and randomization assessment, the patient will be informed to which group he belongs and he will be responsible for scheduling the next maintenance appointment, according to the group to which he belongs.

The study researcher will be responsible for checking if all participants have planned and carried out their maintenance according to his group. He will make sure that they underwent the catheter maintenance in the recommended time period. The study will consist of two arms, with the control group consisting of patients undergoing catheter care every 60 days as recommended in the current institutional protocol. The experimental group will consist of patients who will have a maintenance every 90 days.

Patients will be followed up for one year, with those randomized to the control group having 6 appointments and the experimental group having 4 appointments, in addition to the recruitment period. During follow-up, nurses responsible for this procedure will evaluate the development of specific mechanical complications related to the catheter. A graduated scale of 1 to 5 will be applied: Grade 1 - no resistance to saline infusion with venous return; Grade 2 - no resistance to saline infusion without venous return; Grade 3 - resistance to saline infusion with venous return; Grade 4 - resistance to saline infusion without venous return; Grade 5 - inability to infuse saline without venous return (obstructed). This rating will be recorded on the puncture procedure form already available in the health sector.

In the patient´s cases that will present obstruction in the totally implanted catheter, they will be forwarded to the emergency service. So, the medical teams will evaluate them to verify any possibility to use tissue plasminogen activator (t-PA). In cases of catheter infection, the patient will follow the institutional routine guide of treatment. The puncture procedure will follow the institutional pattern that was validated with the Hospital Infection Control Service.

1.2. Data assessment This study is expected to enrol 410 patients, 205 in the control group and 205 in the experimental group. This evaluation will be performed using the power test with 80% , significance level of 5%, and a rate of 1.35% in obstruction in the control group based on a retrospective study (8) and 2.0% of obstruction in the experimental group with study margin of 2.5% (14).

There are no studies indicating the obstruction rate for the experimental group, so an estimate was made to find the calculated values. If the volume was not collected in the first few months as planned, recruitment may be extended to the two years of this study, during which time as many patients as possible will be recruited.

In the randomization, sequential allocation will be applied (15). As a confusing variable, will be controlled gender and age. As a tool of randomization, an institutional website will be used https://estatsaude.shinyapps.io/alocacao/.

All patients have "intention to treat" and they will be analyzed in the groups they were in until the end of this study. Patients who have more than one event will be counted in each event of the analysis. After data collection, a descriptive analysis will be made. Then the absolute frequency of distribution and relative for qualitative variables and the main measures such as mean, median, and standard deviation and minimum and maximum for quantitative variables.

In order to evaluate a possible association between two qualitative variables, the independence test ( Chi-Square Test or Fisher's exact test) will be used. To compare quantitative variables concerning two independent groups, a non-parametric test of Mann-Whitney or T-test will be used.

Logistic regression models will be applied to evaluate association with clinical and socioeconomic variables of groups between those who will presented or not will presented obstruction of infection of the catheter. The adopted level of significance will be of 5% and the SPSS® for Windows® program, version 22.0 will be used.

1.3. Expected Results This study aims to demonstrate that saline maintenance every 90 days compared with 60-days maintenance does not result in more obstructions or infections in patients undergoing clinical follow-up.

1.4. Possible limitations of this study

The main limitations of this study are that it is a single center study, recruitment difficulty, and decreasing number of participants during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old
* Consent to participate by signing the consent form.
* No intravenous antineoplastic therapy regimen schedule (clinical follow-up).
* To have a functioning, fully implantable catheter with venous return, no resistance during solution infusion, no obstruction or evidence of infection at the time of recruitment.

Exclusion Criteria:

- Use of any type of anticoagulant / antiplatelet drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter obstruction or catheter-related infection | 1 year
  This evaluation will be performed using the power test with 80% , significance level of 5%, and a rate of 1.35% in obstruction in the control group based on a retrospective study (8) and 2.0% of obstruction in the experimental group with study margin of 2.5%

SECONDARY OUTCOMES:
Financial toxicity | 1 year
  Identifying the impact of the economic burden associated with central catheter maintenance with compare groups. The questionnaire has six questions and was produced by the researcher. It will be identified: Work situation (working or not), cost of food, transport, and time on the maintenance day. In addition to the form of health cost (insurance or private)

CONTACTS AND LOCATIONS:
Overall Officials: José Luiz Gasparini-Jr, RN, MSc, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- A.C.Camargo Cancer Center, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No